CLINICAL TRIAL: NCT05317767
Title: Double-blind, Comparative, Randomized Tolerability, Safety and Immunogenicity Trial of Flu-M [Inactivated Split Influenza Vaccine], vs. the Ultrix® Vaccine in Children Aged 6 to 17 Years (Inclusive)
Brief Title: The Objectives of This Study Are Comparative Assessment of the Tolerability, Safety and Immunogenicity of the Flu-M Vaccine vs. the Ultrix® Vaccine by Single Vaccination of Children Aged 6 to 17 Years.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: St. Petersburg Research Institute of Vaccines and Sera (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: FLU-III-D-07/19
Record Dates: First submitted 2021-10-26; First posted 2022-04-08 (Actual); Last update posted 2022-04-08 (Actual); Status verified 2021-10

CONDITIONS: Influenza
Keywords: influenza; flu; vaccine; Flu-M; FluM; Ultrix; SPbSRIVS
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Flu-M (Experimental): 300 children that will be vaccinated with a single dose of the Flu-M vaccine intramuscularly at a dose of 0.5 mL (150 children aged 12 to 17 years, 150 children aged 6 to 11 years)
  Interventions: Biological: Flu-M [Inactivated split influenza vaccine]
- Ultrix (Active Comparator): 300 children that will be vaccinated with a single dose of the Ultrix® vaccine intramuscularly at a dose of 0.5 mL (150 children aged 12 to 17 years, 150 children aged 6 to 11 years)
  Interventions: Biological: Inactivated Split Influenza Vaccine

INTERVENTIONS:
Biological: Flu-M [Inactivated split influenza vaccine] — solution for intramuscular injection, 0.5 ml
  Arms: Flu-M
Biological: Inactivated Split Influenza Vaccine — solution for intramuscular injection, 0.5 ml
  Arms: Ultrix

SUMMARY:
Comparative assessment of the tolerability, safety and immunogenicity of the Flu-M vaccine vs. the Ultrix® vaccine by single vaccination of children aged 6 to 17 years.

DETAILED DESCRIPTION:
At Stage I of the trial, it is planned to screen not more than 350 children aged 12 to 17 years (12 years 0 months 0 days - 17 years 11 months 30 days), of which it is planned to include and randomize 300 children meeting the inclusion and non-inclusion criteria.

Based on findings from tolerability and safety assessment in respect of the Flu-M vaccine vs. the Ultrix® vaccine in the first 7 days after the vaccination of volunteers, during Phase I, an "Opinion on Tolerability and Safety Assessment for the Flu-M Vaccine vs. the Ultrix® Vaccine Involving Children Aged 12-17 Years (12 Years 0 Months 0 Days - 17 Years 11 Months 30 Days) will be prepared/

During Phase II , the trial for Phase I volunteers will continue in full in accordance with the Clinical Trial Regulations.

During the trial, not more than 350 children aged between 6 - 11 years (6 years 0 months - 0 days - 11 years 11 months 30 days) will be further screened, of which it is planned to include and randomize 300 children meeting the inclusion criteria and not falling under the non-inclusion criteria.

ELIGIBILITY:
Inclusion Criteria:

For volunteers aged 12 to 17 years:

* Healthy children1 of both sexes aged 12 to 17 years (12 years 0 months 0 days - 17 years 11 months 30 days);
* The written and dated informed consent of the volunteer (children aged 14-17 years) one of the parents for participation in the trial;
* If the volunteer has sexual relations, effective contraception methods must be used during the 30 days preceding vaccination and consent must be obtained to continue using these contraceptive methods during the trial and for two months after vaccination;
* The girls with mensis in the medical history shall have a negative pregnancy test result.

For volunteers aged 6 to 11 years:

* Healthy children of both sexes aged 6 to 11 years (6 years 0 months 0 days - 11 years 11 months 30 days);
* The written and dated informed consent of one of the parents for participation in the trial;

For all volunteers:

• Ability of a volunteer / volunteer's parents to fulfill the requirements of the Protocol (i.e. to fill out the Patient Diary, come to visit with the volunteer)

Exclusion Criteria:

History of influenza or previous influenza vaccination during 6 months before the trial;

* Vaccination with any vaccine less than 30 days before participating in the trial or scheduled vaccination with any vaccine within 30 days after vaccination with the trial vaccines;
* A serious post-vaccination reaction (temperature above 40 °C, hyperemia or edema more than 8 cm in diameter) or complications (collapse or shock-like condition that developed within 48 hours after vaccination; convulsions accompanied or not accompanied by a fever due to any previous vaccination);
* Allergic reactions to vaccine components or any previous vaccination;
* History of allergic reaction to chicken protein;
* Encephalopathy that developed within 7 days of a previous vaccine administration;
* History of hematopoietic system, cancer;
* Carriage of HIV, syphilis, hepatitis B and C in the medical history, including by parents;
* Children who received immunoglobulin products or transfusions of whole blood or its components less than 3 months before the start of the trial;
* Long-term use (for more than 14 days) of any immunomodulating drugs (immunoregulating peptides, cytokines, interferons, immune system effector proteins (immunoglobulins), interferon inducers (cycloferon)) less than 3 months prior to the commencement of the trial;
* Any confirmed or suspected immunosuppressive or immunodeficiency condition;
* History of chronic diseases of the cardiovascular, bronchopulmonary, endocrine systems, blood in the acute stage (recovery less than 4 weeks before vaccination) or in the decompensation stage;
* History of progressive neurological pathology, convulsive syndrome, afebrile convulsions;
* Acute infectious or non-infectious diseases less than 2 weeks before vaccination;
* Participation in another clinical trial less than 3 months before the start of the trial;
* Smoking (for children of older age group);
* Drug or alcohol abuse in the medical history (for children of older age group);
* Serious concurrent illnesses or pathological conditions not listed above which, in the opinion of the investigator, could complicate the assessment of the results of the trial including pathological deviations from age norms and norms of laboratory blood and urine parameters, which are clinically significant in the opinion of the investigator, or which may be a counter-indicative to participation in the trial in the opinion of the investigator;
* History of mental illness of the volunteer's parents

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 600 (Actual)
Dates: Start 2020-02-10 (Actual); Primary Completion 2020-07-05 (Actual); Study Completion 2020-09-14 (Actual)

PRIMARY OUTCOMES:
Change from Baseline Geometric mean antibodies titer (GMT) at 28 days | Days 0-28
Change from Baseline Seroconversion rate at 28 days | Days 0-28
  An increase in the geometric mean titers of antibodies at Day 28 vs. the baseline level, expressed in the fold rise.
  Seroconversion level ≥ 40%.
Change from Baseline Seroprotection rate at 28 days | Days 0-28
  The percentage of subjects with a generated protective influenza haemagglutinin antibody titer (HA titer) (at least 1:40) vs. the baseline level.
  Seroprotection level ≥ 70%.
Change from Baseline Seroconversion factor at 28 days | Days 0-28
  The percentage of subjects who have a prevaccination titer of HA titer <1:10 and a post-vaccination HA titer >1:40 OR a prevaccination HA titer > 1:10 and at least a fourfold increase in post-vaccination HA titer vs. the baseline.
  Seroconversion factor ≥ 2.5.

SECONDARY OUTCOMES:
Immediate adverse events | During 2 hours after vaccination
  Allergic reactions that revaccination and are reported either by a volunteer / volunteer's parents to the clinical investigator
Adverse events | During 7 days after vaccination
  Local or systemic reactions that are reported either by a clinical investigator or by a volunteer / vaccinated volunteer's parents by phone
Incidence of severe adverse events during the trial | Measurements will be taken then up to 28 days post-vaccination

CONTACTS AND LOCATIONS:
Locations (2):
- Russia (2):
  - Perm State Medical University named after Academician E. A. Wagner, Perm
  - LLC "Meditsinskie Tehnologii", Saint Petersburg